CLINICAL TRIAL: NCT01777659
Title: Transcutaneous Electrical Nerve Stimulation Improves Vascular Conductance After Coronary Artery Bypass Graft Surgery
Acronym: TEBCABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: University of Brasilia (Other); Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, GASPAR ROGERIO DA SILVA CHIAPPA, Principal Investigator, Dr, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-0317
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Acute Myocardial Infarction
Keywords: exercise; neuromodulation; blood flow; exercise capacity
MeSH Terms: conditions — Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS CABG (Experimental): Eligible patients will be randomized to a transcutaneous electrical nerve stimulation program (TENS; n = 20) or to placebo-TENS (P-TENS; n = 18). All patients were followed by their own physicians, received routine nursing assistance, and were visited daily by one of the investigators, but P-TENS group will be not exposed to any specific electrical stimulation or motor physical intervention.
  Interventions: Device: Transcutaneous electrical nerve stimulation
- P-TENS CABG (Placebo Comparator): Patients will be treated with placebo-TENS (P-TENS) condition for 5 days (4 times/day; 30 min/session) applied on cervical region (C7-T4). P-TENS device underwent modifications in its internal programming: the control capacitor of the time constant was changed and the active time between pulses was modified from 330 milliseconds to 33 seconds, in order to prevent an analgesic effect (33).
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — Patients will be treated with conventional TENS (ENDOMED 684 Device, ENRAF-Nonius B.V., Rotterdam, Netherlands) for 5 days (4 times/day; 30 min/session) applied on cervical region (C7-T4). TENS intervention was applied as described elsewhere.
  Other Names: TENS; electrical stimulation

SUMMARY:
The investigators will test the hypothesis that transcutaneous electrical nerve stimulation (TENS) may attenuate peripheral vasoconstriction and to improve blood flow redistribution during handgrip exercise in acute myocardial infarction (AMI) patients after Coronary Arterial Bypass Graft Surgery (CABG).

DETAILED DESCRIPTION:
Thirty-eight patients will be randomized to a (4 times/day; 30 min/session) for 5-day program of TENS (n = 20) or to placebo-TENS (P-TENS, n = 18) applied on cervical region (C7-T4). Acute sympathetic stimulation by cold pressor test (CPT), Maximal voluntary contraction (MVC), Femoral blood flow (FBF) and femoral vascular conductance (FVC) will be measured as primary outcome pre and post-CABG, even as the 6-minute walk test (6-MWT), Inspiratory and expiratory muscle strength (PImax and PEmax) and β-endorphin as a secondary clinical parameters. In addition, amount of opioid analgesic and pain intensity also will be measured throughout at first 24 hours after CABG (immediately, 6, 12 and 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* a previous history of more than 1 vessel coronary artery disease,
* lifelong abstinence from tobacco, and
* formal indication for CABG, according to established guideline.

Exclusion Criteria:

* Patients older than 70 years of age, with chronic renal failure, or with unstable angina in the 48 h prior to CABG, moderate or severe valve disease, complex cardiac arrhythmias, stroke, and/or inability to exercise the lower limbs.

Ages: 48 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Blood flow redistribution - baseline and 5 days later | 1 day
  The ultrasound Doppler system will be equipped with two linear array transducers operating at an imaging frequency of 7- 8 megahertz (MHz). The common femoral artery of the left leg will be insonated distal to the inguinal ligament, 2-3 cm proximal to the bifurcation. Using femoral artery diameter and mean blood velocity (MBF), femoral blood flow (FBF) was calculated as MBF π x (vessel diameter/2)2 x 60. Femoral vascular resistance (FVR) and femoral vascular conductance (FVC) were calculated as (MBP/FBF) and (FBF/MBP * 100 mm Hg), the conductance multiplied by 100 mmHg so that the conductance units will be similar to the units of femoral blood flow (10, 45). The magnitude of reduction FVC (expressed in %) was calculated as vascular conductance during exercise (% change) - conductance at rest (% change) expressed by % of baseline.

SECONDARY OUTCOMES:
Inspiratory and Expiratory Muscle Function | 5 day
  Inspiratory and expiratory muscle strength testing were performed using a pressure transducer (MVD-500 V.1.1 Micro Hard System, Global Med, Porto Alegre, Brazil). Maximal inspiratory (PImax), and maximal static expiratory pressure (PEmax) were measured as previously described.

OTHER OUTCOMES:
Pain Intensity | 5 day
  A visual analog scale (VAS) for assessing current pain intensity will be used to evaluate pain from 0 to 10, where 0 means no pain and 10 indicates severe pain, being applied on the first and on the 5th day after CABG .
Opioid Analgesic Amount | 5 day
  During the first 24 h (immediately, 6, 12 and 24 h) after CABG, the amount of additional analgesic dose (pethidine hydrochloride (HCl) 20 mg, maximum 1 mg/kg/day) was measured for patients in both groups.
β-Endorphin Analysis | 5 day
  Ten milliliters of venous blood will be taken by the phlebotomist. 3 ml of which will be stored in ethylenediaminetetraacetic acid (EDTA) for analysis of a differential white cell count. Seven ml of blood will be divided between an EDTA tube and a lithium heparin (LH) gel tube. These blood samples will be centrifuged and frozen until assayed. β-endorphin was measured by sandwich enzyme immunoassay (ELISA) kit (Phoenix Pharmaceuticals, Inc., USA).

CONTACTS AND LOCATIONS:
Overall Officials: Gaspar R Chiappa, Dr, ScD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil